CLINICAL TRIAL: NCT02201355
Title: A Phase I Study of Reduced-Volume Hypofractionated, PET-directed Intensity Modulated Radiotherapy Concurrent With Weekly Cisplatin Chemotherapy for T1/2N0-2 Squamous Cell Carcinoma of the Head and Neck
Brief Title: Hypofractionated Reduced-Volume Chemoradiation for T1/2N0-2 SCC Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI LEFT THE DEPARTMENT
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 112013-007
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck T1/2N0-2
Keywords: Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemoradiation (Experimental): Hypofractionated, PET-directed, Intensity Modulated Radiotherapy Concurrent with Weekly Cisplatin Chemotherapy
  Interventions: Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy — Patients treated five fractions per week with radiotherapy dose per fraction and cisplatin dose increased according to the treatment table
  Other Names: Hypofractionated,

SUMMARY:
Primary Objectives:

To determine whether patients with T1/2N0-2 Squamous Cell Carcinoma of the oropharynx, hypopharynx or larynx can tolerate treatment with cisplatin chemoradiation in three weeks using reduced volume IMRT

Secondary Objectives:

To describe the adverse events associated with hypofractionated, reduced volume cisplatin chemoradiation.

To estimate response rates and progression-free survival rates of hypofractionated, reduced volume cisplatin chemoradiation.

To determine HRQOL following hypofractionated, reduced volume cisplatin chemoradiation.

If patients can safely be treated in three weeks rather than six weeks, such a schedule would provide a much more convenient alternative for patients and result in a significant reduction in the health care resources currently expended on cure of these patients.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinomas (HNSCC) are frequently occurring tumors with more than 500,000 new cases worldwide and 45,000 in the USA yearly . Most patients present with local-regionally advanced diseases. Chemotherapy given concurrently with radiation is an integrated treatment component in the management of these patients. Concurrent chemoradiation can be given in unresectable diseases, in organ preservation to avoid surgery and preserve functions, and in high risk patients after surgery . Randomized clinical trials and meta-analyses have shown that concurrent chemoradiation are superior to radiation alone in these settings.

One way of reducing overall treatment time and toxicity is to reduce the number of fractions by increasing the daily radiotherapy dose. The consequence of increased daily dose is both an increase in acute side effects as well as an increase in late toxicity. A widely accepted model of these radiobiologic effects over the range of typical 2-4 Gy daily fractions is the alpha-beta model that distinguishes acute responses and late responses based on a linear-quadratic fitting of extrapolated clonogenic survival curves. A time factor can be incorporated to account for the effect of repopulation. Equivalent biologically effective dose schedules using a reduced number of fractions may be calculated for any conventionally fractionated course. Because 70Gy/35/6 weeks with chemoradiation has been demonstrated to be tolerable, and because 66Gy/30/6 weeks has been shown with IMRT to produce 90% control for T1/2 oropharyngeal primary tumors, we will take the biological equivalent of 66Gy/33 fractions over six weeks as the biologic equivalent standard we wish to maintain in hypofractionated courses of radiation. Because 54Gy/30 over six weeks is a well-known elective radiation dose schedule producing 95% control of occult nodal disease, we will take this as the biologically equivalent standard we wish to maintain in our hypofractionated schedules.

ELIGIBILITY:
Inclusion Criteria:

1. T1/2N0-2M0 SCC of the oropharynx, hypopharynx or larynx
2. Age ≥ 18 years.
3. Performance status ECOG 0-1
4. Adequate organ and marrow function as determined by medical oncology evaluation.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

6. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  7 Ability to understand and the willingness to sign a written informed consent.

  8. Creatinine clearance (CC) ≥ 50 ml/min within 4 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)]/[(Serum Cr mg/dl) x (72)] (CCr female = 0.85 x (CrCl male)).

  9. History/physical examination within 4 weeks prior to registration, including assessment of weight and weight loss in past 6 months.

  10. Medical oncology examination to evaluate medical contraindications prior to start chemotherapy 11 Dental evaluation with management prior to start of radiation 12 Nutrition evaluation with consideration of percutaneous endoscopic gastrostomy (PEG) tube placement 13 No distant metastasis by PET/CT

Exclusion Criteria:

1. T3/4 or N3
2. T1N0 disease
3. Metastatic disease
4. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
6. Primary site of tumor of oral cavity, nasopharynx, sinuses, or salivary glands
7. Neck adenopathy that involves the overlying skin.
8. Initial surgical treatment including tonsillectomy or neck dissection, but excluding diagnostic biopsy of the primary site or nodal sampling of neck disease
9. Pre-existing grade > 2 peripheral sensory neuropathy
10. Subjects may not be receiving any other investigational agents.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Treatment completion | 3 weeks
  To determine whether patients with locally advanced SCC of the oropharynx, hypopharynx or larynx can tolerate treatment with cisplatin chemoradiation in three weeks using reduced volume IMRT.

SECONDARY OUTCOMES:
adverse events | 90 days
  To describe the adverse events associated with hypofractionated, reduced volume cisplatin chemoradiation.
progression-free survival rates | 5 years
  To estimate response rates and progression-free survival rates of hypofractionated, reduced volume cisplatin chemoradiation.
Health-related quality of life | 2 years
  To determine HRQOL following hypofractionated, reduced volume cisplatin chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Lucien Nedzi, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas at Southwestern Medical Center, Dallas, Texas, United States